CLINICAL TRIAL: NCT03530397
Title: A Phase 1, Open-label, Dose-escalation and Dose-expansion Study to Evaluate the Safety, Tolerability Pharmacokinetics Immunogenicity, and Antitumor Activity of MEDI5752 in Subjects With Advanced Solid Tumors.
Brief Title: A Study to Evaluate MEDI5752 in Subjects With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D7980C00001; 2018-003075-35 (EudraCT Number)
Record Dates: First submitted 2018-03-28; First posted 2018-05-21 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Selected Advanced Solid Tumors
Keywords: Advanced solid tumors; MEDI5752; immuno-oncology; Cancer; PD-1/CTLA-4 Bispecific; PD-1; CTLA-4; Bispecific; Chemotherapy; Pemetrexed; Carboplatin; Pembrolizumab
MeSH Terms: conditions — Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Pemetrexed; Carboplatin; pembrolizumab; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: MEDI5752 (Experimental): MEDI5752
  Interventions: Biological: MEDI5752
- Arm B: MEDI5752 and chemotherapy (Experimental): MEDI5752, pemetrexed, carboplatin and paclitaxel.
  Interventions: Biological: MEDI5752; Drug: Pemetrexed; Drug: Carboplatin; Drug: Paclitaxel or Nab-Paclitaxel
- Arm C: Pembrolizumab and chemotherapy (Active Comparator): pembrolizumab, pemetrexed, and carboplatin
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Biological: Pembrolizumab

INTERVENTIONS:
Biological: MEDI5752 — Subjects will remain on treatment until unacceptable toxicity, documentation of progressive disease, or development of other reason for treatment discontinuation.
  Arms: Arm A: MEDI5752; Arm B: MEDI5752 and chemotherapy
Drug: Pemetrexed — Subjects will remain on treatment until unacceptable toxicity, documentation of progressive disease, or development of other reason for treatment discontinuation
  Arms: Arm B: MEDI5752 and chemotherapy; Arm C: Pembrolizumab and chemotherapy
Drug: Carboplatin — Subjects will remain on treatment until unacceptable toxicity, documentation of progressive disease, or development of other reason for treatment discontinuation
  Arms: Arm B: MEDI5752 and chemotherapy; Arm C: Pembrolizumab and chemotherapy
Biological: Pembrolizumab — Subjects will remain on treatment until unacceptable toxicity, documentation of progressive disease, or development of other reason for treatment discontinuation
  Arms: Arm C: Pembrolizumab and chemotherapy
Drug: Paclitaxel or Nab-Paclitaxel — Subjects will remain on treatment until unacceptable toxicity, documentation of progressive disease, or development of other reason for treatment discontinuation
  Arms: Arm B: MEDI5752 and chemotherapy

SUMMARY:
The purpose of this study is to evaluate MEDI5752 and carboplatin and pemetrexed or paclitaxel or nab-paclitaxel in adult subjects with advanced solid tumors, when administered as a single agent or combined with chemotherapy.

DETAILED DESCRIPTION:
This is a phase 1, first-time-in-human, multicenter, open-label, dose-escalation and dose-expansion study to evaluate the safety and tolerability, and efficacy, pharmacokinetics and Immunogenicity of MEDI5752 and carboplatin and pemetrexed or paclitaxel or nab-paclitaxel in adult subjects with advanced solid tumors, when administered as a single agent or combined with chemotherapy.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years at the time of screening
2. World Health Organization/Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment
3. Life expectancy ≥ 12 weeks
4. Histologically or cytologically-confirmed advanced solid tumors
5. Subjects who have received prior anti-PD-1, anti-PD-L1, or anti-CTLA-4 therapy or any concurrent chemotherapy, radiotherapy, investigational, biologic, or hormonal therapy for cancer treatment may be eligible to enter the study following a washout period as applicable
6. Females of childbearing potential who are sexually active with a nonsterilized male partner must use at least one highly effective method of contraception
7. Nonsterilized males who are sexually active with a female partner of childbearing potential must use a male condom with spermicide where locally available from Day 1 and for 90 days after the final dose of investigational product. Males receiving pemetrexed or carboplatin must use contraception during study treatment and up to 6 months thereafter.
8. Subjects must have at least one measurable lesion
9. Adequate organ and marrow function
10. Written informed consent and any locally required authorization
11. Subjects must provide tumor material as applicable

Exclusion Criteria

1. Involvement in the planning and/or conduct of the study (applies to both MedImmune staff and/or staff at the study site)
2. Concurrent enrollment in another clinical study, unless it is an observational clinical study or the follow-up period of an interventional study
3. For subjects who have received prior anti-PD-1, anti-PD-L1, or anti-CTLA-4:

   1. Subjects must not have received anti-PD-1, anti-PD-L1, anti-CTLA-4 or any other immunotherapy or immune-oncology (IO) agent within 21 days of commencing treatment with investigational product.
   2. Subject must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
   3. All AEs while receiving prior immunotherapy must have completely resolved or resolved to Grade 1 prior to screening for this study.
4. Current or prior use of immunosuppressive medication within 14 days before the first dose of investigational product is excluded.
5. Receipt of live attenuated vaccine within 30 days prior to the first dose of investigational product.
6. Active or prior documented autoimmune or inflammatory disorders
7. History of active primary immunodeficiency:
8. History of organ transplant
9. Known allergy or reaction to any component of the planned study treatment.
10. Untreated CNS metastatic disease, leptomeningeal disease, or cord compression
11. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v4.03 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria
12. Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of Investigational Product or still recovering from prior surgery
13. Female subjects who are pregnant or breastfeeding, as well as male or female subjects of reproductive potential who are not willing to employ one highly effective method of birth control
14. Uncontrolled intercurrent illness, that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the subject to give written informed consent.
15. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of the subject's safety or study results
16. Judgment by the investigator that the subject is unsuitable to participate in the study and the subject is unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The number of subjects experiencing treatment related adverse events (AEs) (Dose-escalation phase) | From the time of informed consent through 114 days following termination of treatment with investigational product
  The primary endpoint is as assessed by the number of subjects experiencing adverse events (AEs) graded per NCI CTCAE v4.03
Preliminary anti-tumor activitiy of MEDI5752 (versus pembrolizumab, where applicable) using Objective Response based on RECIST v1.1 (Dose-expansion phase) | From the first dose of study drug through the date of first documented progression, end of study, date of death, or two years after the last patient starts treatment, whichever should occur first
  The primary endpoint of antitumor activity include Objective Response and will be based on all post baseline disease assessments that occur prior to initiation of subsequent anticancer therapy.
The number of subjects experiencing dose-limiting toxicities (DLTs) (Dose-escalation phase) | Up to 21 days following the first dose
  The primary endpoint is as assessed by the number of subjects experiencing dose limiting toxicities (DLTs) as defined by the protocol.
The number of subjects experiencing abnormal laboratory evaluations (Dose-escalation phase) | From the time of informed consent through 114 days following termination of treatment with investigational product
  The primary endpoint is as assessed as the number of subjects experiencing changes in laboratory parameters from baseline.
The number of subjects experiencing changes from baseline in vital signs reported as adverse events (Dose-escalation phase) | From the time of informed consent through 114 days following termination of treatment with investigational product
  The primary endpoint is as assessed by the number of subjects experiencing clinically significant changes in vital signs from baseline.
The number of subjects experiencing abnormal electrocardiograms (ECG) reported as Adverse Events (Dose-escalation phase) | From the time of informed consent through 114 days following termination of treatment with investigational product
  The primary endpoint is as assessed by the the number of subjects experiencing clinically significant changes in ECG parameters from baseline.
The number of subjects experiencing treatment related serious adverse events (SAEs) (Dose-escalation phase) | From the time of informed consent through 114 days following termination of treatment with investigational product
  The primary endpoint is as assessed by the number of subjects with serious adverse events (SAEs) graded per NCI CTCAE v4.03.

SECONDARY OUTCOMES:
Pharmacokinetics of MEDI5752: Cmax | To be assessed at Day 1, 2, 3, 8, 15, 22, 29, 43, 64, 85, and 106 over the first 4 months of treatment and up to 114 days following end of treatment
  The endpoints for the assessment of PK of MEDI5752 include individual MEDI5752 concentrations at different time points after administration. PK parameters that may be modeled on this data include maximum observed concentration (Cmax)
Pharmacokinetics of MEDI5752: AUC | To be assessed at Day 1, 2, 3, 8, 15, 22, 29, 43, 64, 85, and 106 over the first 4 months of treatment and up to 114 days following end of treatment
  The endpoints for the assessment of PK of MEDI5752 include individual MEDI5752 concentrations at different time points after administration. PK parameters that may be modeled on this data include area under the concentration-time curve (AUC)
Pharmacokinetics of MEDI5752: Clearance | To be assessed at Day 1, 2, 3, 8, 15, 22, 29, 43, 64, 85, and 106 over the first 4 months of treatment and up to 114 days following end of treatment
  The endpoints for the assessment of PK of MEDI5752 include individual MEDI5752 concentrations at different time points after administration. PK parameters that may be modeled on this data include clearance (CL)
Pharmacokinetics of MEDI5752: t 1/2 | To be assessed at Day 1, 2, 3, 8, 15, 22, 29, 43, 64, 85, and 106 over the first 4 months of treatment and up to 114 days following end of treatment.
  The endpoints for the assessment of PK of MEDI5752 include individual MEDI5752 concentrations at different time points after administration. PK parameters that may be modeled on this data include terminal phase half life (t 1/2)
Ability of MEDI5752 to generate immune response in subjects with advanced solid tumors | To be assessed at Day 1, 8, 15, 22, 29, 43, 64, 85, and 106 over the first 4 months of treatment and up to 114 days following end of treatment.
  The endpoints for the immunogenicity of MEDI5752 include the number of subjects who develop detectable anti-drug antibodies (ADAs)
PD-L1 Expression in subjects with advanced solid tumors | To be assessed at baseline
  The endpoint for the PD-L1 expression will be determined by Immunohistochemistry characterization.
Preliminary Antitumor Activity: Duration of Response | From the date of response through the date of first documented progression, end of study, date of death, or two years after last subject starts treatment whichever should occur first
  The endpoints for assessment of antitumor activity include duration of response (DoR) and is defined as the duration from the documentation of OR to the first documentation of disease progression or death due to any cause.
Preliminary Antitumor Activity: Disease Control | From the first dose of study drug through the date of first documented progression, end of study, date of death, or two years after last subject starts treatment whichever should occur first
  The endpoints for assessment of antitumor activity include disease control (DC) and is defined as CR, PR, or SD according to RECIST v1.1.
Preliminary Antitumor Activity: Progression Free Survival | From the first dose of study drug through the date of first documented progression, end of study, date of death, or two years after last subject starts treatment whichever should occur first
  The endpoints for assessment of antitumor activity include progression free survival (PFS) and is defined as the duration measured from the start of treatment with investigational product to the first documentation of disease progression or death due to any cause.
Preliminary Antitumor Activity: Overall Survival | From the first dose of study drug through the end of study, or date of death, or two years after last subject starts treatment whichever should occur first
  The endpoints for assessment of antitumor activity include overall survival (OS) and is defined as the duration measured from the start of treatment with investigational product until death due to any cause.
The number of subjects experiencing treatment related adverse events (AEs) (Dose-expansion phase) | From the time of informed consent through 114 days following termination of treatment with investigational product
  The secondary endpoint is as assessed by the number of subjects experiencing adverse events (AEs) graded per NCI CTCAE v4.03
The number of subjects experiencing abnormal laboratory evaluations (Dose-expansion phase) | From the time of informed consent through 114 days following termination of treatment with investigational product
  The secondary endpoint is as assessed by the number of subjects experiencing changes in laboratory parameters from baseline.
The number of subjects experiencing Changes from baseline in vital signs reported as adverse events (Dose-expansion phase) | From the time of informed consent through 114 days following termination of treatment with investigational product
  The secondary endpoint is as assessed by the number of subjects experiencing clinically significant changes in vital signs from baseline.
The number of subjects experiencing abnormal ECGs reported as adverse events (Dose-expansion phase) | From the time of informed consent through 14 days following termination of treatment with investigational product
  The secondary endpoint is as assessed by the number of subjects experiencing clinically significant changes in ECG parameters from baseline.
The number of subjects experiencing treatment related serious adverse events (SAEs) (Dose-expansion phase) | From the time of informed consent through 114 days following termination of treatment with investigational product
  The secondary endpoint is as assessed by the number of subjects with serious adverse events (SAEs) graded per NCI CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Subramaniam, MD, MSc, Principal Investigator — AstraZeneca
Locations (32):
- United States (7):
  - Research Site, Detroit, Michigan
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Providence, Rhode Island
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Fairfax, Virginia
- Australia (2):
  - Research Site, Melbourne
  - Research Site, Randwick
- France (3):
  - Research Site, Bordeaux
  - Research Site, Lyon
  - Research Site, Villejuif
- Italy (4):
  - Research Site, Meldola
  - Research Site, Napoli
  - Research Site, Ravenna
  - Research Site, Roma
- Research Site, Amsterdam, Netherlands
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- South Korea (4):
  - Research Site, Cheongju-si
  - Research Site, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Seoul
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Majadahonda
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Valencia
- Taiwan (3):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home